CLINICAL TRIAL: NCT06346613
Title: Prevalence and Affecting Factors of Sleep and Circadian Rhythm Disorders in ICU: An Observational Study
Brief Title: Prevalence and Affecting Factors of Sleep and Circadian Rhythm Disorders in ICU
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2024-076R
Record Dates: First submitted 2024-03-14; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Sleep Deprivation; Circadian Rhythm Disorders; Critical Illness
Keywords: circadian rhythm; sleep; ICU
MeSH Terms: conditions — Sleep Deprivation; Chronobiology Disorders; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 ml of the patient's blood was drawn and centrifuged to obtain serum, which was used to measure the patient's melatonin levels
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most ICU patients experience sleep and circadian disruption (SCD), which causes a profound negative impact on patients, such as prolonged mechanical ventilation, glucose intolerance, and the occurrence of delirium. In order to better promote the alignment of circadian rhythm in ICU patients, this project will explore the prevalence of SCD and a series of influencing factors contributing to SCD in ICU patients, to help construct targeted intervention programs in the future.

DETAILED DESCRIPTION:
The circadian rhythm refers to the oscillation phenomenon of physiological, biochemical, and behavioral life phenomena of organisms with a 24-hour cycle. The circadian rhythm affects multiple physiological indicators, such as the sleep-wake cycle, hormone levels, heart rate, blood pressure, and metabolic functions. Maintaining a normal circadian rhythm is crucial for human health. However, a series of stressful stressors in the ICU, such as lack of normal light-dark cycle changes, high levels of noise, make sleep and circadian rhythm disruption(SCD) common and severe, and such disruption will have serious negative impacts on patients' clinical outcomes. Therefore, there is an urgent need for effective interventions to assist ICU patients in promoting their sleep and circadian rhythms. The first step in intervention is to understand the current incidence and characteristics of ICU SCD, as well as the factors contributing to such disruption.

To date, there has been limited progress on the current status of SCD prevalence in ICUs. On one hand, there may be significant variability in ICU SCD between individual patients and subgroups, On the other hand, this variability may change over time as patients recover from acute illnesses. This heterogeneity from population and time impedes the development of interventions for SCD. Therefore, there is an urgent need to understand the characteristics, trends of SCD in different patients and the factors influencing these changes.

The overall objective of this project is to explore the status and influencing factors of ICU patients' sleep and circadian rhythms in the first 3 days by conducting a longitudinal study using multiple objective subjective indicators, aiming to more accurately and objectively evaluate the changes in patients' circadian rhythms.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients older than 18 years old.
2. Patients transferred to ICU during the time period of 8:00-22:00.
3. Stay in the ICU for more than 12 hours and at least one overnight period.
4. Patients or their family members are informed and consent to participate in the research.

Exclusion Criteria:

1. Acute brain injuries within 30 days, such as acute intracranial bleeding, traumatic brain injury, central nervous system infection, or chronic brain injuries lasting over 30 days with an inability to live independently.
2. Previously diagnosed with mild cognitive impairment or Alzheimer's disease.
3. Patients affected by blindness or optic nerve disorder.
4. Patients who are pregnant or breastfeeding.
5. Patient in prone position, hemodialysis, or ECMO therapy during PSG monitoring
6. Imminently dying or with a hospice status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the Surgical Intensive Care Unit (SICU) at Zhongshan Hospital, Fudan University, critically ill adult patients from both surgical and medical specialties are admitted in SICU.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rhythmicity of melatonin levels. | Starting from 3:00 on the first day after admission to the ICU, four blood samples are taken every day (at 3:00, 9:00, 15:00, and 21:00), continuing for three days.
  Measuring the patient's circadian rhythm using their melatonin secretion levels.

SECONDARY OUTCOMES:
Overnight sleep duration | During the first three nights after entering the ICU.
  Minutes of sleep from 22:00 to 6:00 as measured by portable polysomnography device (Alice PDX)
Wake after sleep onset(WASO) | During the first three nights after entering the ICU.
  Minutes of WASO from 22:00 to 6:00 as measured by portable polysomnography device (Alice PDX)
Overnight Rapid Eye Movement (REM) proportion | During the first three nights after entering the ICU.
  Proportion of Stage REM sleep from 22:00 to 6:00 as measured by portable polysomnography device (Alice PDX)
Overnight non-rapid eye movement stage 1 (NREM1) proportion | During the first three nights after entering the ICU.
  Proportion of Stage NREM1 sleep from 22:00 to 6:00 as measured by portable polysomnography device (Alice PDX)
Overnight non-rapid eye movement stage 2 (NREM2) proportion | During the first three nights after entering the ICU.
  Proportion of Stage NREM2 sleep from 22:00 to 6:00 as measured by portable polysomnography device (Alice PDX)
Overnight non-rapid eye movement stage 3 (NREM3) proportion | During the first three nights after entering the ICU.
  Proportion of Stage NREM3 sleep from 22:00 to 6:00 as measured by portable polysomnography device (Alice PDX)
Sleep period time ratio (sleep continuity) | During the first three nights after entering the ICU.
  Nighttime sleep duration divided by the number of nighttime sleep cycles, sleep data is measured by portable polysomnography device (Alice PDX) from 22:00 to 6:00.
Subject sleep quality | Within 12 hours after each PSG measurement
  Using the Richards-Campbell Sleep Questionnaire to measure the sleep quality of patients.
Activity counts | Starting from 22:00 on the first day after admission to the ICU, continuing for three days.
  The activity count is recorded by actigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: YuXia Zhang, PhD, Study Director — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guan T, Li J, Hou J, Pan W, Liu X, Cai S, Zhang Y. Prospective cohort study on characteristics, associated factors and short-term prognosis of sleep and circadian rhythm in intensive care unit: protocol for the SYNC study. BMJ Open. 2025 Mar 4;15(3):e091184. doi: 10.1136/bmjopen-2024-091184. PMID 40037668